CLINICAL TRIAL: NCT01443156
Title: The Effects of Work Schedule and Sleep Patterns on Caregivers' Health
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jackilen Shannon, Scientist, Oregon Health and Science University
Other Study IDs: OHSU eIRB7542
Record Dates: First submitted 2011-09-20; First posted 2011-09-29 (Estimated); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Obesity; Diabetes; Cancer; Metabolic Syndrome; Sleep Deprivation
Keywords: Diet; Sleep deficiency; Cancer; Obesity; Diabetes; Shift work; Work schedule; Cardiovascular disease; Body composition; Body mass index; Body fat percentage
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Neoplasms; Metabolic Syndrome; Sleep Deprivation; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Mouthwash swish containing buccal cells.

GROUPS / COHORTS (1):
- Caregivers: Employees at a local medical facility, including (but not limited to): nurses, laboratory technicians, non-clinical hospital staff

SUMMARY:
BACKGROUND. Sleep deficiency (not getting enough sleep) is widespread in American adults and can lead to many harmful health outcomes such as a higher risk of obesity, heart disease, and diabetes. Sleep deficiency can also harm cognitive performance, which refers to one's awareness and thinking ability. Sleep deficiency and sleep-related health issues are of high interest among those who have irregular and/or extended work schedules, because such schedules can interfere with normal biological rhythms of sleepiness and wakefulness.

PURPOSE. This study will examine the health and cognitive effects of work schedule and sleep patterns in caregivers (such as nurses, laboratory technicians, and non-clinical hospital staff). The investigators hypothesize that the nontraditional, irregular, and extended work hours common in these professions will have adverse health and cognitive effects. The purposes of this protocol are to:

* Enroll caregivers into a one year cohort study on the relationships among work schedule, sleep, diet, chronic disease, and cognitive performance. (A cohort study follows a group of participants over time to see how different behaviors or risk factors affect health.)
* Collect data from caregivers on work schedule, sleep, diet, chronic disease, and cognitive performance.
* Give personalized information and feedback to caregivers about these health factors.
* Educate caregivers about healthy diet and exercise choices.
* Collect saliva from caregivers for future research on the role of genes in health. (Specimen collection for genetic testing will be offered as a separate option for study participants.) RECRUITMENT. This study will use the Let's Get Healthy! health research and education program (OHSU IRB #3694) as a platform for recruitment and data collection. Caregivers will be invited to participate in a Let's Get Healthy! event and will be given information prior to the event about the cohort study. At the Let's Get Healthy! event, caregivers will first consent to the anonymous research study (OHSU IRB #3694), in which demographic and health screening data are linked to a random number. Caregivers will then have the option to consent to a cohort study, in which data are no longer anonymous but instead linked to participants' names and contact information.

PROCEDURES. This cohort study piggybacks on procedures already approved for the Let's Get Healthy! program (OHSU IRB #3694). Let's Get Healthy! is a study in which participants provide anonymous data at health fairs through any or all of the following manners: short computer surveys on cancer awareness, risk factors, and family history (with immediate feedback given on cancer risk and prevention); short computer surveys on diet and sleep patterns (with immediate printed feedback given); health screening measurements (blood pressure, height, weight, waist circumference, body mass index, body fat percentage); a finger stick to assess sugar and fat levels in blood; and a mouthwash swish to provide a saliva specimen.

However, this cohort study (OHSU IRB #7542) will make the following changes and additions:

* Personal health data, instead of being anonymous, will be linked to participants' names and contact information (for follow-up data collection).
* Let's Get Healthy! events will include cognitive performance tests, a preventative-care survey, and a work schedule survey.
* Participants will provide data not only at an initial Let's Get Healthy! event, but also at a follow-up event and during the time period between events. Between events, participants will do the surveys on work schedule, diet, and sleep, and they will complete cognitive performance tests.
* There will be a separate consent process for participants to provide a fully identifiable saliva specimen.

DATA ANALYSIS. Participants' health data will be fully identifiable at the time of data collection but will be coded and stored in a physically separate location from the identifiable information. The link between identifiable information and coded health information will be stored on a password protected computer, and all identifiable information will be deleted upon completion of data analyses. Data will be analyzed to explore relationships among work schedule, sleep, diet, body composition, metabolic health, chronic disease, and cognitive performance in caregivers. Genetic relationships with these factors will be analyzed in those who provided a saliva specimen during entry visit data collection.

ELIGIBILITY:
Inclusion Criteria:

* Employed caregiver in a hospital setting
* 18 years of age or older
* Completion of minimal set of stations (see below, section III.d.)
* Consent given electronically

Exclusion Criteria:

* Declining to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cohort participants will be recruited from employees at a local health care center. Job categories may include, but are not limited to:
  * Administrative services
  * Clinical services (radiology, laboratory, pharmacy, etc.)
  * Clinical support services (aide, clerk, processing, records, etc.)
  * Practitioner (physician, physician assistant, nurse practitioner, etc.)
  * Non-clinical services (food, nutrition, housekeeping, etc.)
  * Nursing services-registered nurse
  * Nursing services-certified nursing assistant
  * Rehabilitative services (occupational therapy, speech therapy, physical therapy, etc.)
Sampling Method: Non-Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2012-01; Primary Completion 2013-02 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Cognitive performance | Up to one year
  Brief computerized tasks of attention, vigilance, and memory.
Body Composition | Up to one year
  Height, weight, waist circumference, body fat percentage, body mass index
Diet | Up to one year
  Brief computerized survey on fruit, vegetable, and fat intake.
Work Schedule | Up to one year
  Survey on the quantity and distribution of work hours.

SECONDARY OUTCOMES:
Blood Pressure | Up to one year
Blood cholesterol, glucose, triglycerides | Up to one year
  Fingerstick test
Breast, skin, and lung cancer prevention behaviors and knowledge | Up to one year
  Brief computerized questionnaires.
Preventive care habits | Up to one year
  Brief survey on basic health behaviors and use of preventive care resources.

CONTACTS AND LOCATIONS:
Overall Officials: Jackilen Shannon, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- St. Charles Medical Center, Bend, Oregon, United States